CLINICAL TRIAL: NCT02725086
Title: Evaluation of Pharmacokinetic/Pharmacodynamic Properties and Safety of Leucostim® Compared to Neupogen® in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DA3030_NP_I
Record Dates: First submitted 2016-03-22; First posted 2016-03-31 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
MeSH Terms: interventions — Filgrastim

ARMS (2):
- Part 1; Filgrastim 5 ㎍/kg (Experimental): Neupogen®(Filgrastim) 5 ㎍/kg or Leucostim®(Filgrastim) 5 ㎍/kg will be administered subcutaneously on Period 1, Day 1. And wash out for 28 days or more. Leucostim®(Filgrastim) 5 ㎍/kg or Neupogen®(Filgrastim) 5 ㎍/kg will be administered subcutaneously on Period 2, Day 1.
  Interventions: Drug: Leucostim®; Drug: Neupogen®
- Part 2; Filgrastim 10 ㎍/kg (Experimental): Neupogen®(Filgrastim) 10 ㎍/kg or Leucostim®(Filgrastim) 10 ㎍/kg will be administered subcutaneously on Period 1, Day 1. And wash out for 28 days or more. Leucostim®(Filgrastim) 10 ㎍/kg or Neupogen®(Filgrastim) 10 ㎍/kg will be administered subcutaneously on Period 2, Day 1.
  Interventions: Drug: Leucostim®; Drug: Neupogen®

INTERVENTIONS:
Drug: Leucostim®
  Other Names: DA-3030
Drug: Neupogen®

SUMMARY:
A Randomized, Open-label, Two-way Crossover, Open-label Clinical Trial to Compare Pharmacokinetic/Pharmacodynamic Properties and Safety after Subcutaneous Administration of Leucostim® and Neupogen® in Healthy Adult Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Age 19 - 45 years
* BMI 18.5 - 25.0 kg/m2
* Value of ANC(absolute neutrophil count) had to be inside the normality range at the screening

Exclusion Criteria:

* Subjects with a history or presence of clinically relevant hypersensitivity reaction to investigational drugs (G-CSF) or their ingredients/additives
* Subjects with a clinically relevant history of allergic reaction
* Subjects with a history of acute infectious diseases within 2 weeks prior to administration of investigational products
* At the investigator's discretion, subjects who is considered inappropriate to participate in the study due to any conditions including screening results

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
AUCinf of Filgrastim | 0~48 hr
  PK parameter
Cmax of Filgrastim | 0~48 hr
  PK parameter
AUEC0-t of ANC(absolute neutrophil count) | 0~120 hr
  PD parameter
Emax of ANC(absolute neutrophil count) | 0~120 hr
  PD parameter

SECONDARY OUTCOMES:
Tmax of Filgrastim | 0~48 hr
  PK parameter
AUC0-t of Filgrastim | 0~48 hr
  PK parameter
CL/F of Filgrastim | 0~48 hr
  PK parameter
Vd/F of Filgrastim | 0~48 hr
  PD parameter
AUEC0-t of CD34+ cell count | 0~312 hr
  PD parameter
Emax of CD34+ cell count | 0~312 hr
  PD parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University College of Medicine, Seoul, Seodamun-gu, South Korea